CLINICAL TRIAL: NCT00226681
Title: Nursing Interventions Following Sudden Cardiac Arrest
Brief Title: Nurses Helping Sudden Cardiac Arrest Survivors Recover After Getting An Implantable Cardioverter Defibrillator (ICD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Cynthia M. Dougherty ARNP, PhD, University of Washington; Biobehavioral Nursing & Health Systems
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 4766; R01NR004766 (NIH)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Nursing Telephone Support Protocol
- 2 (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Nursing Telephone Support Protocol
  Arms: 1
Behavioral: Usual Care
  Arms: 2

SUMMARY:
To determine if an education and support nursing intervention program helped sudden cardiac arrest survivors adjust to the event and to getting an ICD

DETAILED DESCRIPTION:
This study is one of the first large randomized clinical trials of nursing interventions aimed at improving health outcomes after receiving an ICD. Written informed consent was used in the study.

ELIGIBILITY:
Inclusion Criteria:

* First time sudden cardiac arrest with ICD implantation during hospitalization, over age 21 years, working telephone in the home, deliverable address for 1 year

Exclusion Criteria:

* Receiving an ICD for primary prevention of sudden cardiac arrest, inability to read, speak, or understand English, no telephone at home or no current address, cognitive or physical impairments that prohibited ability to give informed consent.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1999-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To determine if an education and support nursing intervention program helped sudden cardiac arrest survivors adjust to the event and to getting an ICD | Baseline, 1- and 3-months from implantation

SECONDARY OUTCOMES:
Improved physical functioning | Baseline, 1- and 3-months from implantation
Improved psychological adjustment | Baseline, 1- and 3-months from implantation
Improved self-efficacy | Baseline, 1- and 3-months from implantation
Lower health care use | Baseline, 1- and 3-months from implantation

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Dougherty, ARNP, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Dougherty CM, Lewis FM, Thompson EA, Baer JD, Kim W. Short-term efficacy of a telephone intervention by expert nurses after an implantable cardioverter defibrillator. Pacing Clin Electrophysiol. 2004 Dec;27(12):1594-602. doi: 10.1111/j.1540-8159.2004.00691.x. PMID 15613121